CLINICAL TRIAL: NCT04523883
Title: Randomized Phase II Trial of Postoperative Radiotherapy With Concurrent JS001（PD-1 Antibody） vs. Postoperative Radiotherapy Alone in Intermediate/High-risk Head and Neck Cancer Patients With a Contraindication to Cisplatin
Brief Title: Concurrent Immunotherapy With Postoperative Radiotherapy in Intermediate/High Risk HNSCC Patients Unfit for Cisplatin: The IMPORT Study (IMPORT)
Acronym: IMPORT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Collaborators: Fudan University (Other); Eye & ENT Hospital of Fudan University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); First Affiliated Hospital of Fujian Medical University (Other); Guizhou Provincial People's Hospital (Other); Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020HNRT03
Record Dates: First submitted 2020-08-18; First posted 2020-08-24 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-08

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; radiotherapy; PD-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concurrent PD-1 (Experimental): Concurrent Immunotherapy With Postoperative Radiotherapy
  Interventions: Radiation: postoperative radiotherapy; Drug: JS001
- Radiotherapy alone (Active Comparator): Postoperative Radiotherapy alone
  Interventions: Radiation: postoperative radiotherapy

INTERVENTIONS:
Radiation: postoperative radiotherapy — postoperative radiotherapy with a dose of 60-66Gy
Drug: JS001 — JS001 240mg every three week
  Other Names: Toripalimab
  Arms: concurrent PD-1

SUMMARY:
To investigate weather concurrent JS001 with postoperative radiotherapy would have survival benefit in intermediate/high Risk HNSCC Patients who cannot take cisplatin

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologically confirmed squamous cell carcinoma of the head and neck.Site of tumor origin in the oral cavity, oropharynx, larynx, hypopharynx , or sinuses (excluding nasopharynx) 2. With at least one risk factors after radical surgery ①positive margin; ②close margin（<5mm); ③ENE;④PNI;⑤LVI; ⑤ pT3-4/N2-3( AJCC 8th).⑥ Level IV/V lymph node metastases for OPC or OC.

  3. Have at least one contraindication to cisplatin as defined:

  ① Age>65 years old; ②Creatinine clearance (CC) > 30 and < 60 cc/min For this calculation, use the Cockroft-Gault formula: CC = 0.85 (if female)* ((140-Age) / (Serum Creatinine)) * (Weight in kg / 72); ③ Zubrod performance status 2; ④Pre-existing peripheral neuropathy grade ≥ 1; ⑤History of hearing loss, defined as either: ▪ Existing need of a hearing aid OR ≥ 25 decibel shift over 2 contiguous frequencies on a pretreatment hearing test as clinically indicated.

  4. No distant metastases 5. No synchronous or concurrent head and neck primary tumors 6. ECOG PS 0-2 7. Adequate organ function including the following:
  1. Absolute neutrophil count (ANC) >= 1.5 * 10^9/l
  2. Platelets count >= 80 * 10^9/l
  3. Hemoglobin >= 80 g/dl
  4. AST and ALT <= 2.5 times institutional upper limit of normal (ULN)
  5. Total bilirubin <= 1.5 times institutional ULN
  6. Creatinine clearance >30 ml/min 8. Signed written informed consent

Exclusion Criteria:

1. Prior chemotherapy or anti-cancer biologic therapy for any type of cancer, or prior radiotherapy to the head and neck region
2. Other previous cancer, except for in situ cervical cancer and cutaneous basal cell carcinoma
3. Pregnant or breast-feeding females, or females and males of childbearing potential not taking adequate contraceptive measures
4. Uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia
5. Active, known or suspected autoimmune disease such as interstitial pneumonia, uveitis, Crohn's disease, autoimmune thyroiditis. Subjects with cured childhood asthma, type I diabetes mellitus and hypothyroidism only requiring hormone replacement, or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment
6. Using systemic immunosuppressive agents and continue the dose within 2 weeks prior to the enrollment;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-08-09 (Estimated); Study Completion 2024-08-09 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | from date of enrollment until date of first documented disease progression or death from any cause, assessed up to 2 years

SECONDARY OUTCOMES:
Overall survival | from date of enrollment until death from any cause, assessed up to 2 years
Number of participants with treatment-related acute toxicity as assessed weekly by CTCAE v4.0 during the course of treatment | up to 3 months after completion of radiotherapy
  Acute toxicity profiles, graded according to the NCI CTCAE version 4.0
Number of participants with treatment-related late toxicity as assessed by CTCAE v4.0 | from 3 months after completion of radiotherapy up to 2 years
  Late toxicity profiles, graded according to the NCI CTCAE version 4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Guopei Zhu, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided